CLINICAL TRIAL: NCT00455065
Title: Weight Loss and Cardiovascular Disease (CVD) Prevention Via a Whole Grain Diet in Men and Women With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB20474
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome
Keywords: whole grain; metabolic syndrome; weight loss
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Whole Grain Foods

SUMMARY:
The purpose of this study is to determine if intake of whole grain foods as part of a hypocaloric diet enhances weight loss and improves cardiovascular disease risk factors in men and women with metabolic syndrome.

DETAILED DESCRIPTION:
Fifty men and women with metabolic syndrome age 20 to 65 will be recruited to participate. Men and women are eligible if they have a body mass index (BMI) ≥ 30 and at least three out of five ATP III criteria for metabolic syndrome. These criteria are defined as: [1] Triacylglycerol ≥150 mg/dL, [2] HDL <40 mg/dL in men or <50 mg/dL in women, [3] Fasting glucose ≥100 mg/dL, [4] Systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥85 mg/dL, and [5] waist circumference ≥102 cm in men or ≥88 cm in women.

Participants will receive dietary advice to either avoid whole grain foods or to have all of their grain servings each day from whole grain foods for 12 weeks. Participants will be stratified by gender and BMI and randomized using a random number table. A registered dietitian will meet individually with each participant at baseline to discuss the dietary intervention and provide educational materials. Participants in the whole grain group are given a target number of daily whole grain servings, either 4, 5, 6 or 7 servings/d, based on the number of grain servings recommended in the 2005 Dietary Guidelines For Americans for their energy needls to facilitate understanding and adherence. Participants in the whole grain group are given a list and description of whole grain foods to help them identify foods to include in their diet and were encouraged to select foods that had a whole grain food listed as the first ingredient. To ease the transition, participants in the whole grain group will consume three servings of whole grain foods per day for the first two weeks of the study and then increase to their target number of daily whole grain servings for the remaining ten weeks. Participants in the refined grain group are also given a list of whole grain foods and asked not to consume any of these foods during the study period.

In addition to the instruction on whole grain servings, participants in both groups are aasked to eat five servings of fruit and vegetables, three servings of low-fat dairy products, and two servings of lean meat, fish or poultry/d, as recommended in the 2005 Dietary Guidelines for Americans. The target macronutrient composition for all participants is 55% carbohydrate, 30% fat, with emphasis on unsaturated fats, and 15% protein. All participants are encouraged to engage in moderate physical activity at least three times a week for 30 minutes per session and were instructed to avoid dietary supplements throughout the study period. Participants in both groups are told that their aim was to lose at least 1 pound per week for the duration of the study.

Every other week, participants visit the study site and review their diet records with a dietitian on a one-on-one basis. During this time, the dietitian presents an educational lesson that explained the rationale for the dietary guidelines used in the study, and offered nutritional guidance, encouragement, and suggestions for improvement. The participant's weight, blood pressure, and waist circumference are also recorded. On the weeks that participants do not come in for a study visit, they are contacted by phone or e-mail by a dietitian to discuss their progress and address any concerns or questions. A fasting blood draw, 2-hour oral glucose tolerance test (OGTT), dual energy x-ray absorptiometery (DXA) scan, and biometric measurements are done at the beginning and end of the 12-week diet period at The Pennsylvania State University General Clinical Research Center (GCRC).

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥ 30
* at least three out of five ATP III criteria for metabolic syndrome. These criteria are defined as: [1] Triacylglycerol ≥150 mg/dL, [2] HDL <40 mg/dL in men or <50 mg/dL in women, [3] Fasting glucose ≥100 mg/dL, [4] Systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥85 mg/dL, and [5] waist circumference ≥102 cm in men or ≥88 cm in women.

Exclusion Criteria:

* diagnosis of type I or II diabetes
* diagnosis of CVD
* diagnosis of cancer
* diagnosis of any other serious medical condition
* use of any medications that affect glucose, insulin, cholesterol, or reproductive hormones
* smoker
* drink more than 2 alcoholic beverages/d
* consume a diet high in whole grains (>3 servings/d)
* pregnant or lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Weight Loss

SECONDARY OUTCOMES:
Waist Circumference
Blood Pressure
Body fat percentage
Lipids and Lipoproteins
Glucose Tolerance (OGTT)
Testosterone Concentration
Markers of Inflammation and Fibrinolysis

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, Ph.D., Principal Investigator — Penn State University

REFERENCES:
- [Derived] Katcher HI, Legro RS, Kunselman AR, Gillies PJ, Demers LM, Bagshaw DM, Kris-Etherton PM. The effects of a whole grain-enriched hypocaloric diet on cardiovascular disease risk factors in men and women with metabolic syndrome. Am J Clin Nutr. 2008 Jan;87(1):79-90. doi: 10.1093/ajcn/87.1.79. PMID 18175740